CLINICAL TRIAL: NCT05836103
Title: Testing the Impact of Smartphone-based Messaging to Support Young Adult Smoking Cessation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00013413
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Tobacco Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: The investigators propose to test tailored smartphone-based messages to support young adults in quitting smoking. This study addresses 3 specific aims.
  For Aim 1, a micro-randomized trial (within-subject randomization) with 80 young adult smokers will investigate the efficacy of smoking cessation messages based on CBT and mindfulness/ACT for reducing smoking urge 15 minutes after message delivery.
  In Aim 2, a built-in and conventionally randomized EMA-only control group will allow us to test if intervention messages result in changes in smoking behavior over time. The primary outcome will be self-reported number of cigarettes per day at end of treatment, as well as 3- and 6-month follow-up.
  Aim 3 will explore moderation effects of substance co-use (cannabis, alcohol, other drugs) and exposure to specific locations (home, work, bars) on urge reduction message efficacy among intervention group participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micro-randomized trial group (Experimental): The micro-randomized trial will determine if CBT and Mindfulness/ACT messages are superior to control messages in reducing the primary outcome momentary smoking urges. Based on participants' training data collected in the initial 14 days of EMA monitoring, intervention messages will be delivered during time-periods and at high-risk locations for smoking. In the intervention phase, participants will be prompted to complete 3 geofence-triggered EMAs per day for a total of 30 days. Each EMA will be followed by an intervention message and the type of message (CBT, Mindfulness/ACT, control) will be randomly selected at each time point (within-subject randomization).
  Interventions: Behavioral: Smartphone-based intervention messages
- EMA-only control group (No Intervention): A total of N=80 participants will be randomized into an EMA-only control group, parallel to the micro-randomized trial intervention group. This group will conduct 14-day EMA only training phase just like the micro-randomized trial group, but will not be switched over to the intervention phase after these initial 14 days. Instead, participants will continue the EMA-only data collection procedure for an additional 30-days (analogous to the 30-day intervention phase of the micro-randomized trial). During these 30 days, the EMA-only control group will continue to receive 3 randomly prompted EMA surveys per day and an additional 3 EMA surveys triggered by smoking reports.

INTERVENTIONS:
Behavioral: Smartphone-based intervention messages — Intervention messages in the proposed trial will address specific high-risk situations for smoking and smoking urges. Messages will focus on two key situational triggers for message matching: 1. Stress (high/low) and 2. Presence of other smokers (yes/no). For each situation, characterized by a combination of these characteristics, several messages were developed. To improve user engagement with the intervention, all messages contain visual content in form of pictures.
  Arms: Micro-randomized trial group

SUMMARY:
Clinical practice guidelines for smoking cessation emphasize cognitive behavioral therapy (CBT) to help patients develop coping strategies for urges. Mindfulness or Acceptance and Commitment Therapy (ACT) offer a different approach, which teaches smokers psychological flexibility through accepting negative experiences. While there is evidence for the efficacy of both CBT and Mindfulness/ACT smoking cessation interventions, it is unclear if these approaches are efficacious when implemented in real-time and with young adults. The overall goal of this proposal is to evaluate the efficacy of CBT and Mindfulness/ACT messages for young adults targeted at specific high-risk situations for smoking.

DETAILED DESCRIPTION:
This research will address the following specific aims:

Aim 1: To test CBT and Mindfulness/ACT intervention message efficacy for reducing momentary smoking urges (N=80). To inform just-in-time interventions, it is crucial to test if CBT and Mindfulness/ACT based messages can reduce momentary smoking urges. The investigators will conduct a micro-randomized trial (repeated within-subject randomizations of messages) to accomplish this. In line with the investigators' existing protocol, participants first collect Ecological Momentary Assessment (EMA) data for 14 days, allowing the investigators to determine high-risk situations for smoking. In the following intervention phase, participants receive tailored messages triggered by geofencing of participants' high-risk locations for a total of 30 days. Tailoring is based on established predictors of smoking relapse (stress and presence of other smokers). The micro-randomized trial tests the efficacy of CBT versus Mindfulness/ACT versus control messages for reducing smoking urge 15 minutes post message delivery. Secondary outcomes include smoking or other tobacco use (including e-cigarettes), affect, and stress.

Aim 2: To test if exposure to urge reduction messages results in changes in smoking behavior over time compared to an EMA only control group (N=80). It is important to investigate if repeated messages in the micro-randomized trial impact smoking behavior over time, in contrast to just repeated assessment without messages. Thus, this study includes a conventionally randomized clinical-trial component. Parallel to the micro-randomized trial group, a control group completes EMA surveys only without intervention messages. This allows the investigators to test if messages reduce smoking behavior. The primary outcome is number of cigarettes per day at end of treatment, 3-, and 6-months follow-up. Secondary analyses explore biochemically verified 7-day point prevalence abstinence, switching to e-cigarettes, and other tobacco outcomes. Post-hoc dose-response analyses investigate the long-term efficacy of CBT or Mindfulness/ACT messages on smoking behavior.

Aim 3: Explore moderation effects of substance co-use (cannabis, alcohol, other drugs) and exposure to specific location (home, work, bars) on urge reduction message efficacy. A crucial research question to inform future mobile interventions is how well intervention messages work in different situational contexts and when people are co-using other substances. Among intervention group participants, the investigators will explore how urge reduction message efficacy may be moderated by substance co-use and exposure to specific settings.

ELIGIBILITY:
Inclusion Criteria:

1. live in the U.S.
2. read English;
3. are between 18 and 30 years of age;
4. own an iPhone or Android smartphone;
5. have smoked ≥100 cigarettes in their lives and currently smoke at least 3 cigarettes per day on 5 or more days of the week;
6. are planning to quit smoking within the next 30 days.

Exclusion Criteria:

* None

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in smoking urge as assessed by a single item | 15 minutes after message delivery
  The primary outcome will be change in participants' rating of smoking urge in EMA-post surveys, prompted 15 minutes after intervention message delivery, and controlling for the ratings in EMA-pre surveys. Urge will be assessed by a single item on a 5-point scale, ranging from 1 (very low) to 5 (very high).
Change in cigarettes smoked per day in past week as assessed by a single item | Baseline, 45-day, 3-month, and 6-month follow-up
  The primary outcome will be change in self-reported number of cigarettes smoked per day in the past week from baseline to 45-day, 3-month, and 6-month follow-up.

SECONDARY OUTCOMES:
Smoking since intervention message delivery as assessed by a single item | 15 minutes after message deliery
  Smoking in the 15 minutes after message delivery will be assessed by a single item on a binary response scale (yes/no).
Other tobacco product use since intervention message delivery as assessed by a single item | 15 minutes after message delivery
  Other tobacco product use, including e-cigarette use, in the 15 minutes after message delivery will be assessed by a single item on a binary response scale (yes/no).
Change in stress as assessed by a single item | 15 minutes after message delivery
  Change in rating of stress in EMA-post surveys, prompted 15 minutes after intervention message delivery, and controlling for the ratings in EMA-pre surveys. Stress will be assessed by a single item on a 5-point scale, ranging from 1 (very low) to 5 (very high).
Change in negative affect as assessed by a single item | 15 minutes after message delivery
  Change in rating of negative affect in EMA-post surveys, prompted 15 minutes after intervention message delivery, and controlling for the ratings in EMA-pre surveys. Negative affect will be assessed by a single item on a 5-point scale, ranging from 1 (very low) to 5 (very high).
Message helpfulness as assessed by a single item | 15 minutes after message delivery
  Rating of message helpfulness in EMA-post surveys, prompted 15 minutes after intervention message delivery. This will be assessed by a single item on a 5-point scale, ranging from 1 (not at all helpful) to 5 (extremely helpful).
Activity completion as assessed by a single item | 15 minutes after message delivery
  Self-reported completion of intervention message recommendation in EMA-post surveys, prompted 15 minutes after intervention message delivery will be assessed by a single item on a binary response scale (yes/no).
Self-reported 7-day point prevalence abstinence as assessed by a single item | 45-day follow-up
  Self-reported 7-day point prevalence abstinence (no smoking, not even a puff) will be assessed by a single item on a binary response scale (yes/no).
Self-reported 7-day point prevalence abstinence as assessed by a single item | 3-month follow-up
  Self-reported 7-day point prevalence abstinence (no smoking, not even a puff) will be assessed by a single item on a binary response scale (yes/no).
Self-reported 7-day point prevalence abstinence as assessed by a single item | 6-month follow-up
  Self-reported 7-day point prevalence abstinence (no smoking, not even a puff) will be assessed by a single item on a binary response scale (yes/no).
Saliva-cotinine confirmed 7-day point prevalence abstinence | 45-day follow-up
  Saliva-cotinine confirmed 7-day point prevalence abstinence. This will be assessed using saliva test strips and photo confirmation.
Saliva-cotinine confirmed 7-day point prevalence abstinence | 3-month follow-up
  Saliva-cotinine confirmed 7-day point prevalence abstinence. This will be assessed using saliva test strips and photo confirmation.
Saliva-cotinine confirmed 7-day point prevalence abstinence | 6-month follow-up
  Saliva-cotinine confirmed 7-day point prevalence abstinence. This will be assessed using saliva test strips and photo confirmation.
Change in cigarettes smoked as assessed by a single item | Baseline, 45-day, 3-month, and 6-month follow-up
  Change (reduction) in cigarettes smoked by at least 50% between baseline and each follow-up timepoint. Reduction will be calculated based on self-reported number of cigarettes/day in the past week.
Tobacco quit attempt as a assessed by a single item | Baseline, 45-day, 3-month, and 6-month follow-up
  A tobacco quit attempt since last assessment will be assessed by a single item on a binary response scale (yes/no).
Change in frequency and intensity of smoking urges as assessed by two items of the Mood and Physical Symptoms Scale (MPSS) | Baseline, 45-day, 3-month, and 6-month follow-up
  Change in frequency and intensity of smoking urges will be assessed by two craving items from the Assessed with the Mood and Physical Symptoms Scale (MPSS) - subscale MPSS(C). Both items will be assessed on a 6-point scale from 0 (not at all / no urges) to 5 (all the time / extremely strong). Both items will be combined into the MPSS(C) subscale for analysis.
Change in psychological flexibility as assessed by the CompACT-15 | Baseline, 45-day, 3-month, and 6-month follow-up
  Change in psychological flexibility from baseline to 45-day, 3-month, and 6-month follow-up will be assessed by the CompACT-15. The CompACT-15 total score ranges from 0-90, with higher scores indicating greater psychological flexibility.
Change in smoking-specific experiential avoidance as assessed by the Avoidance and Inflexibility Scale (AIS) | Baseline, 45-day, 3-month, and 6-month follow-up
  Change in smoking-specific experiential avoidance from baseline to 45-day, 3-month, and 6-month follow-up will be assessed by the Avoidance and Inflexibility Scale (AIS). Items are scored on a scale of 1-5 and combined into a total score. A higher total score indicates a more avoidant and inflexible response to internal states associated with smoking.
Tobacco product switching as assessed by 5 questions | Baseline, 45-day, 3-month, and 6-month follow-up
  Switching to other tobacco products including e-cigarettes from baseline to 45-day, 3-month, and 6-month follow-up will be assessed using questions about past 7-day use of cigarettes, e-cigarettes, cigars / cigarillos / little cigars, smokeless tobacco, and hookah / waterpipe. Participants will be coded as having switched if they do not report cigarette smoking, but use of another tobacco product at a follow-up assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Thrul, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Any individual requests for data will be honored on a case-by-case basis as deemed appropriate to the research protocol.
Supporting Information: Study Protocol, Analytic Code

REFERENCES:
- [Derived] Thrul J, Devkota J, Waring JJC, Desjardins MR, Hamoud J, Han J, Naughton F, Zipunnikov V, Mendelson T, Latkin C, Epstein D, Moran M. App-Based Smoking Urge Reduction Intervention for Young Adults: Protocol Combining a Microrandomized Trial and Conventional Between-Subject Randomized Trial. JMIR Res Protoc. 2025 Sep 23;14:e74388. doi: 10.2196/74388. PMID 40987452